CLINICAL TRIAL: NCT02387372
Title: A Phase 1, Prospective, Multi-center, Open-label Study to Assess the Plasma Pharmacokinetics and Lung Penetration of Intravenous (IV) Ceftolozane/Tazobactam in Critically Ill Patients
Brief Title: Plasma Pharmacokinetics (PK) & Lung Penetration of Ceftolozane/Tazobactam in Participants With Pneumonia (MK-7625A-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7625A-007; CXA-ICU-14-01 (Other: Cubist Pharmaceuticals LLC Protocol Number)
Record Dates: First submitted 2015-01-12; First posted 2015-03-13 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Critically Ill; Pneumonia
MeSH Terms: conditions — Critical Illness; Pneumonia | interventions — ceftolozane; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanically Ventilated (Experimental): Participants with proven or suspected pneumonia, undergoing mechanical ventilation will receive 4-6 doses of ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion as follows:
  * Those with Creatinine clearance (CLCR) > 50 mL/min will receive 4-6 doses of 3 g ceftolozane/tazobactam every 8 hours
  * Those with CLCR 30 - 50 mL/min will receive 4-6 doses of 1.5 g ceftolozane/tazobactam every 8 hours
  * Those with CLCR 15 - 29 mL/min will receive 6 doses of 750 mg ceftolozane/tazobactam every 8 hours
  Interventions: Drug: Ceftolozane/Tazobactam - Multiple Doses
- Critically Ill (Experimental): Critically ill participants with CLCR ≥180 mL/min (as calculated by the Cockcroft-Gault equation) will receive a single dose of ceftolozane/tazobactam, 3 g, as a 60-minute intravenous infusion.
  Interventions: Drug: Ceftolozane/Tazobactam - Single Dose

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam - Multiple Doses — 4-6 doses of ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion as follows:
  * Participants with CLCR > 50 mL/min will receive 4-6 doses of 3 g ceftolozane/tazobactam every 8 hours
  * Participants with CLCR 30 - 50 mL/min will receive 4-6 doses of 1.5 g ceftolozane/tazobactam every 8 hours
  * Participants with CLCR 15 - 29 mL/min will receive 6 doses of 750 mg ceftolozane/tazobactam every 8 hours
  Arms: Mechanically Ventilated
Drug: Ceftolozane/Tazobactam - Single Dose — Single dose of ceftolozane/tazobactam, 3 g, as a 60-minute intravenous infusion
  Arms: Critically Ill

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and lung penetration of intravenous Ceftolozane/tazobactam in critically ill participants.

DETAILED DESCRIPTION:
This is a Phase 1, prospective, multicenter, non-comparative, open-label study to characterize the plasma pharmacokinetics and intrapulmonary penetration of ceftolozane/tazobactam in two groups of participants.

Group 1: approximately 25 ventilated participants with suspected or proven pneumonia receiving concurrent standard antibiotic therapy. Within Group 1, efforts will be made to enroll approximately 5 participants with a CLCR ≥ 150 mL/min (as calculated by the Cockcroft-Gault equation).

Group 2: 8-10 critically ill participants with CLCR ≥180 mL/min (as calculated by the Cockcroft-Gault equation).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study-related procedure not part of normal medical care.
2. If female,must not be pregnant or nursing, and is either:

   1. Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or
   2. Of childbearing potential and:

      * Is practicing an effective method of contraception (e.g., oral/parenteral contraceptives or a barrier method) and for at least 1 month prior to baseline assessments, or
      * Has a vasectomized partner, or
      * Is currently abstinent from sexual intercourse. Participants must be willing to practice the chosen contraceptive method or remain abstinent during the conduct of the study and for at least 30 days after last dose of study medication.
3. Non-vasectomized males are required to practice effective birth control methods (e.g., abstinence, use of a condom or use of other barrier device) during the conduct of the study and for at least 30 days after last dose of study medication;
4. Participants in Group 1 must meet the following criteria:

   1. Males or females age 18 years or older;
   2. Intubated and on mechanical ventilation for at least 24 hours prior to time of enrollment (includes participants with tracheostomy who are mechanically ventilated);
   3. Proven or suspected bacterial pneumonia, as confirmed by the presence of at least one of the prescribed clinical signs and symptoms.
   4. Receiving antibiotic therapy for proven or suspected bacterial pneumonia at the time of enrollment and expected to continue on antibiotic therapy while in the study
5. Participants in Group 2 must meet the following criteria:

   1. Males or females aged 18 - 54 years;
   2. Acute Physiology and Chronic Health Evaluation II (APACHE II) score between 12 and 35, inclusive;
   3. CLCR ≥180 mL/min (as calculated by the Cockcroft-Gault equation using actual body weight) within 24 hours of dosing;
   4. Documented infection or presumed infection.

Exclusion Criteria:

1. Has a documented history of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibacterial (a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment);
2. Hemoglobin < 7 g/dL at baseline;
3. Prior (within 24 hours of first dose of study drug) or concomitant receipt of piperacillin/tazobactam, probenecid or ceftolozane/tazobactam (non-study use);
4. Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the Investigator);
5. Any condition or circumstance that, in the opinion of the Investigator, would compromise the safety of the participant or the quality of study data;
6. Planned or prior participation in any interventional drug study within the last 30 days;
7. Participants in Group 1 must not meet any of the following criteria:

   1. Receipt of effective systemic antibiotic therapy for the treatment of proven or suspected bacterial pneumonia for more than 72 hours prior to start of the first dose of study drug
   2. Any of the following diagnoses or conditions that may interfere with the PK assessment/interpretation:

      * Cystic fibrosis, acute exacerbation of chronic bronchitis or obstructive airway disease, chronic severe respiratory disease , or active pulmonary tuberculosis,
      * Full thickness burns (greater than 15% of total body surface area),
      * Lung transplant recipient or donor,
      * Any condition or situation where bronchoscopy is not advisable;
8. End-stage renal disease defined as a CLCR < 15 mL/min (as calculated by the Cockcroft-Gault equation using actual body weight), OR requirement for continuous renal replacement therapy or hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Nicolau DP, De Waele J, Kuti JL, Caro L, Larson KB, Yu B, Gadzicki E, Zeng Z, Rhee EG, Rizk ML. Pharmacokinetics and Pharmacodynamics of Ceftolozane/Tazobactam in Critically Ill Patients With Augmented Renal Clearance. Int J Antimicrob Agents. 2021 Apr;57(4):106299. doi: 10.1016/j.ijantimicag.2021.106299. Epub 2021 Feb 7. PMID 33567333
- [Derived] Caro L, Nicolau DP, De Waele JJ, Kuti JL, Larson KB, Gadzicki E, Yu B, Zeng Z, Adedoyin A, Rhee EG. Lung penetration, bronchopulmonary pharmacokinetic/pharmacodynamic profile and safety of 3 g of ceftolozane/tazobactam administered to ventilated, critically ill patients with pneumonia. J Antimicrob Chemother. 2020 Jun 1;75(6):1546-1553. doi: 10.1093/jac/dkaa049. PMID 32211756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult males or non-pregnant or non-nursing females that were mechanically ventilated or critically ill were enrolled in this study.
Period: Overall Study
Arm/Group | Mechanically Ventilated | Critically Ill
Started | 27 | 10
Treated | 26 | 10
Completed | 26 | 10
Not Completed | 1 | 0
Not completed — Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Mechanically Ventilated | Critically Ill | Total
Number analyzed (Participants) | 26 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (15.85) | 36.2 (9.65) | 55.9 (18.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 16 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 23 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 19 | 9 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for creatinine clearance (CLCR), every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Cmax, maximum plasma concentration, of ceftolozane or tazobactam. Pharmacokinetic (PK) data analysis was performed by non-compartmental analysis (NCA) method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: All mechanically ventilated participants who received at least 1 dose of study drug at the correctly assigned dose level, and whose plasma drug concentration was determined. Critically ill participants were not analyzed in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Groups:
- Mechanically Ventilated- Ceftolozane; Mechanically Ventilated -Tazobactam: Participants with proven or suspected pneumonia, undergoing mechanical ventilation will receive 4-6 doses of ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion as follows:
  * Those with Creatinine clearance (CLCR) > 50 mL/min will receive 4-6 doses of 3 g ceftolozane/tazobactam every 8 hours
  * Those with CLCR 30 - 50 mL/min will receive 4-6 doses of 1.5 g ceftolozane/tazobactam every 8 hours
  * Those with CLCR 15 - 29 mL/min will receive 6 doses of 750 mg ceftolozane/tazobactam every 8 hours
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
ug/mL
  First Dose | 73.0 [61.4 to 86.9] | 22.6 [18.9 to 27.1]
  Last Dose: number analyzed (Participants) | 24 | 24
  Last Dose | 100 [84.2 to 120] | 26.1 [21.8 to 31.3]
Statistical Analysis 1: Comparison: Mechanically Ventilated- Ceftolozane; Accumulation Ratio of Last Dose/First Dose; Test type: Other; Geometric least squares mean ratio (GMR) = 1.38, 90% CI 2-sided [1.21 to 1.56] — Ratio of Last Dose/First Dose
Statistical Analysis 2: Comparison: Mechanically Ventilated -Tazobactam; Accumulation Ratio of Last Dose/First Dose; Test type: Other; GMR = 1.15, 90% CI 2-sided [1.03 to 1.29] — Ratio of Last Dose/First Dose

2. Primary Outcome: Epithelial Lining Fluid (ELF) / Plasma Ratio (Intrapulmonary Penetration) of Ceftolozane and Tazobactam Concentrations in Mechanically Ventilated Participants.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples and epithelial lining fluid (ELF) were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the epithelial lining fluid, ELF to plasma ratio of ceftolozane and tazobactam.
Time Frame: Up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of the last infusion.
Population: All mechanically ventilated participants who received at least 1 dose of study drug at the correctly assigned dose level, and whose plasma and ELF drug concentrations were both determined. Critically ill participants were not analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Mechanically Ventilated - Ceftolozane; Mechanically Ventilated - Tazobactam: Participants with proven or suspected pneumonia, undergoing mechanical ventilation will receive 4-6 doses of ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion as follows:
  * Those with Creatinine clearance (CLCR) > 50 mL/min will receive 4-6 doses of 3 g ceftolozane/tazobactam every 8 hours
  * Those with CLCR 30 - 50 mL/min will receive 4-6 doses of 1.5 g ceftolozane/tazobactam every 8 hours
  * Those with CLCR 15 - 29 mL/min will receive 6 doses of 750 mg ceftolozane/tazobactam every 8 hours
Arm/Group | Mechanically Ventilated - Ceftolozane | Mechanically Ventilated - Tazobactam
Number analyzed (Participants) | 22 | 22
Ratio
  1 Hr Post-dose: number analyzed (Participants) | 5 | 5
  1 Hr Post-dose | 0.213 (0.130) | 0.234 (0.140)
  2 Hr Post-dose: number analyzed (Participants) | 5 | 5
  2 Hr Post-dose | 0.360 (0.212) | 0.471 (0.241)
  4 Hr Post-dose: number analyzed (Participants) | 5 | 5
  4 Hr Post-dose | 1.76 (3.24) | 2.34 (4.25)
  6 Hr Post-dose: number analyzed (Participants) | 4 | 4
  6 Hr Post-dose | 1.02 (0.773) | 2.59 (2.36)
  8 Hr Post-dose: number analyzed (Participants) | 3 | 3
  8 Hr Post-dose | 0.786 (0.248) | 1.06 (0.543)

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Tmax, time of maximum plasma concentration, of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
Hours
  First Dose | 1.00 [0.883 to 2.00] | 1.00 [0.883 to 1.12]
  Last Dose: number analyzed (Participants) | 24 | 24
  Last Dose | 1.00 [0.917 to 2.17] | 1.00 [0.917 to 2.17]

4. Primary Outcome: Last Quantifiable Plasma Concentration (Clast) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Clast, last quantifiable plasma concentration, of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
ug/mL
  First Dose | 14.0 [10.3 to 19.0] | 1.14 [0.721 to 1.81]
  Last Dose: number analyzed (Participants) | 24 | 24
  Last Dose | 24.0 [17.7 to 32.5] | 1.52 [0.955 to 2.40]
Statistical Analysis 1: Comparison: Mechanically Ventilated- Ceftolozane; Accumulation Ratio of Last Dose/First Dose; Test type: Other; Geometric least squares mean ratio (GMR) = 1.71, 90% CI 2-sided [1.50 to 1.96] — Ratio of Last Dose/First Dose
Statistical Analysis 2: Comparison: Mechanically Ventilated -Tazobactam; Accumulation Ratio of Last Dose/First Dose; Test type: Other; GMR = 1.33, 90% CI 2-sided [1.14 to 1.55] — Ratio of Last Dose/First Dose

5. Primary Outcome: Time of Last Quantifiable Plasma Concentration (Tlast)) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Tlast, time of last quantifiable plasma concentration, of ceftolozane or tazobactam. PK data analysis was determined by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
Hours
  First Dose | 7.95 [5.77 to 8.17] | 7.95 [5.77 to 8.17]
  Last Dose: number analyzed (Participants) | 24 | 24
  Last Dose | 7.98 [6.12 to 8.33] | 7.98 [6.00 to 8.33]

6. Primary Outcome: Area Under the Concentration Time Curve (AUC) From the First to Time of the Last Dose (AUC0-last) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the AUC0-last, AUC from the first to time of the last dose, of ceftolozane or tazobactam. PK data analysis was determined by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h*ug/mL
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
h*ug/mL
  First Dose | 242 [199 to 293] | 50.7 [40.8 to 63.0]
  Last Dose: number analyzed (Participants) | 24 | 24
  Last Dose | 390 [321 to 473] | 63.0 [50.6 to 78.4]
Statistical Analysis 1: Comparison: Mechanically Ventilated- Ceftolozane; Accumulation Ratio of Last Dose/First Dose; Test type: Other; Geometric least squares mean ratio (GMR) = 1.61, 90% CI 2-sided [1.44 to 1.81] — Ratio of Last Dose/First Dose
Statistical Analysis 2: Comparison: Mechanically Ventilated -Tazobactam; Accumulation Ratio of Last Dose/First Dose; Test type: Other; GMR = 1.24, 90% CI 2-sided [1.11 to 1.39] — Ratio of Last Dose/First Dose

7. Primary Outcome: AUC From the Time of the Dose to Infinity (AUC0-∞) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the AUC0-∞, AUC from the time of the dose to infinity, of ceftolozane or tazobactam. PK data analysis was determined by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h*ug/mL
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
h*ug/mL
  First Dose: number analyzed (Participants) | 24 | 25
  First Dose | 353 [269 to 464] | 58.1 [45.1 to 74.7]
  Last Dose: number analyzed (Participants) | 23 | 23
  Last Dose | 605 [461 to 795] | 69.8 [54.1 to 90.0]
Statistical Analysis 1: Comparison: Mechanically Ventilated- Ceftolozane; Accumulation Ratio of Last Dose/First Dose; Test type: Other; Geometric least squares mean ratio (GMR) = 1.71, 90% CI 2-sided [1.51 to 1.95] — Ratio of Last Dose/First Dose
Statistical Analysis 2: Comparison: Mechanically Ventilated -Tazobactam; Accumulation Ratio of Last Dose/First Dose; Test type: Other; GMR = 1.20, 90% CI 2-sided [1.09 to 1.33] — Ratio of Last Dose/First Dose

8. Primary Outcome: Terminal Elimination Half-life (t1/2) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the t1/2, terminal elimination half-life, of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
Hours
  First Dose: number analyzed (Participants) | 24 | 25
  First Dose | 4.15 (56.1) | 2.15 (56.4)
  Last Dose: number analyzed (Participants) | 23 | 23
  Last Dose | 4.86 (61.5) | 2.33 (49.7)

9. Primary Outcome: Volume of Distribution at Steady State (Vss) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Vss, volume of distribution at steady state, of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
Liter
  First Dose: number analyzed (Participants) | 24 | 25
  First Dose | 27.5 (29.9) | 39.9 (28.9)
  Last Dose: number analyzed (Participants) | 23 | 23
  Last Dose | 29.4 (45.5) | 40.4 (38.8)

10. Primary Outcome: Plasma Clearance (CL) of Ceftolozane or Tazobactam in Mechanically Ventilated Participants for the First and Last Dose of Ceftolozane/Tazobactam Treatment.
Description: Mechanically ventilated participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the CL, plasma clearance, of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 up to Day 2 at 0 (pre-dose), 1, 2, 4, 6 and 8 hours (h) after the start of the first and last infusions.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Mechanically Ventilated- Ceftolozane | Mechanically Ventilated -Tazobactam
Number analyzed (Participants) | 25 | 25
L/h
  First Dose: number analyzed (Participants) | 24 | 25
  First Dose | 4.90 (64.1) | 15.0 (68.5)
  Last Dose: number analyzed (Participants) | 23 | 23
  Last Dose | 4.52 (67.7) | 14.1 (75.6)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 5 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanically Ventilated | Critically Ill
Number analyzed (Participants) | 26 | 10
Participants | 16 | 6

12. Secondary Outcome: Cmax of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Cmax of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: All critically ill participants who received at least 1 dose of study drug at the correctly assigned dose level, and whose plasma drug concentration was determined. Mechanically ventilated participants were not analyzed in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Groups:
- Critically Ill - Ceftolozane; Critically Ill - Tazobactam: Critically ill participants with CLCR ≥180 mL/min (as calculated by the Cockcroft-Gault equation) will receive a single dose of ceftolozane/tazobactam, 3 g, as a 60-minute intravenous infusion.
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 10
ug/mL | 68.9 [55.0 to 86.5] | 17.4 [13.5 to 22.5]

13. Secondary Outcome: Tmax of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Tmax of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 10
Hours | 1.02 [0.983 to 1.07] | 1.02 [0.983 to 1.07]

14. Secondary Outcome: Clast of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Clast of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 10
ug/mL | 5.82 [2.95 to 11.5] | 0.357 [0.153 to 0.833]

15. Secondary Outcome: Tlast of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Tlast of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 10
Hours | 7.95 [7.72 to 8.15] | 7.85 [4.07 to 8.15]

16. Secondary Outcome: AUC0-last of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the AUC0-last of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: h*ug/mL
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 10
h*ug/mL | 188 [139 to 255] | 31.0 [20.3 to 47.5]

17. Secondary Outcome: AUC0-∞ of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the AUC0-∞ of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: h*ug/mL
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 9
h*ug/mL | 233 [152 to 327] | 34.8 [21.7 to 55.9]

18. Secondary Outcome: T1/2 of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the T1/2 of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 9
Hours | 2.59 (51.1) | 1.47 (43.5)

19. Secondary Outcome: Vss of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the Vss of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 9
Liter | 30.2 (41.1) | 51.6 (41.1)

20. Secondary Outcome: CL of Ceftolozane/Tazobactam in Critically Ill Participants With Augmented Renal Function.
Description: Critically ill participants received a 60 minute infusion of ceftolozane/tazobactam, adjusted for CLCR, every 8 hours; then blood samples were collected at 1, 2, 4, 6, and 8 hours post start of the final infusion after the last dose of study drug in order to determine the CL of ceftolozane or tazobactam. PK data analysis was performed by NCA method using Phoenix WinNonlin version 6.3 or later.
Time Frame: Day 1 at 0 (pre-dose), 1, 2, 4, 6 and 8 h after the start of infusion
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Critically Ill - Ceftolozane | Critically Ill - Tazobactam
Number analyzed (Participants) | 10 | 9
L/h | 8.98 (57.6) | 28.7 (67.9)

ADVERSE EVENTS:
Time Frame: Up to 5 days
Description: All treated participants
Groups:
- Mechanically Ventilated: 3 g Ceftolozane/Tazobactam: Participants with proven or suspected pneumonia, undergoing mechanical ventilation received 4-6 doses of 3 g ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion
- Mechanically Ventilated: 1.5 g Ceftolozane/Tazobactam: Participants with proven or suspected pneumonia, undergoing mechanical ventilation received 4-6 doses of 1.5 g ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion
- Mechanically Ventilated: 0.75 g Ceftolozane/Tazobactam: Participants with proven or suspected pneumonia, undergoing mechanical ventilation received 4-6 doses of 0.75 g ceftolozane/tazobactam every 8 hours as a 60-minute intravenous infusion
- Critically Ill: 3 g Ceftolozane/Tazobactam: Critically ill participants with CLCR ≥180 mL/min (as calculated by the Cockcroft-Gault equation) received a single dose of ceftolozane/tazobactam, 3 g, as a 60-minute intravenous infusion.
Arm/Group | Mechanically Ventilated: 3 g Ceftolozane/Tazobactam | Mechanically Ventilated: 1.5 g Ceftolozane/Tazobactam | Mechanically Ventilated: 0.75 g Ceftolozane/Tazobactam | Critically Ill: 3 g Ceftolozane/Tazobactam
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/4 | 0/1 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/4 | 0/1 | 0/10
Other Adverse Events (participants affected / at risk) | 14/21 | 1/4 | 1/1 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mechanically Ventilated: 3 g Ceftolozane/Tazobactam (N=21) | Mechanically Ventilated: 1.5 g Ceftolozane/Tazobactam (N=4) | Mechanically Ventilated: 0.75 g Ceftolozane/Tazobactam (N=1) | Critically Ill: 3 g Ceftolozane/Tazobactam (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT02387372/Prot_SAP_000.pdf